CLINICAL TRIAL: NCT03987399
Title: Pediatric Postoperative Pain Management in Surgical Wards - an Intervention Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Anja Hetland Smeland, Research nurse, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019/388
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Pain
Keywords: pediatric pain; postoperative pain; pain assessment; pain management; healthcare providers; children; nurses; physicians; tailored educational intervention; surgical wards
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tailored educational intervention (Experimental): The intervention will be based on previous research and results from baseline (T1). The intervention will be a one-day educational day and includes lectures and workshops with main focus on the lowest competence in pediatric postoperative pain management. Healthcare providers at the included surgical wards will be invited to participate on this educational day. As a supplement, there will be provided clinical supervision in pediatric postoperative pain management and reminders (such as lectures and posters) over a period of six months after educational day.
  Interventions: Other: Tailored educational intervention

INTERVENTIONS:
Other: Tailored educational intervention — Educational day (lecture and workshop), clinical supervision and reminders

SUMMARY:
This study will explore healthcare providers' pediatric postoperative pain management knowledge and clinical practice. The aim of this study is to explore healthcare providers' knowledge and clinical practice in pediatric postoperative pain management in surgical wards, and to evaluate whether an educational intervention would improve postoperative pain management. This study has a pre-post intervention design. This study will be conducted on four surgical wards in one university hospital in Norway. There will be used different methodological approaches for data collections (interviews, questionnaire, observational study) with four measurement points; baseline (T1), and one month (T2), six months (T3) and 12 months (T4) after intervention.

DETAILED DESCRIPTION:
This study will be conducted on four surgical wards in one university hospital in Norway. There will be used different methodological approaches for data collections (interviews, questionnaire, observational study) with four measurement points; baseline (T1), and one month (T2), six months (T3) and 12 months (T4) after intervention.

To get a broader view of barriers and facilitators for effective pediatric postoperative pain management, there will be carried out focus group interviews with healthcare providers. Further, data about healthcare providers' knowledge and attitudes regarding pediatric pain will be collected using a questionnaire. Data about nurses' pediatric postoperative pain management will be collected using non-participant observational study and data about children's experience about pain and pain management will be collected using face-to-face interviews with children. This study will have different phases:

Phase 1 Explore healthcare providers' knowledge, clinical practice children's experiences of pain and pain management, and healthcare providers' experiences of barriers and facilitators for effective pain management

* Questionnaire PNKAS-N
* Observation of clinical practice
* Face-to-face interviews with children
* Focus group interviews with healthcare providers (barriers and facilitators)

Phase 2 Develop and implement a tailored educational intervention

Develop tailored educational intervention based on:

* Available research
* Results from baseline
* Feedback from head of the relevant units
* Staff views about the facilitators and barriers to optimized pediatric pain management

Implementation of the intervention

* Seminar (lecture and workshop)
* Clinical supervision
* Reminders

Phase 3 Evaluation of the intervention

* Questionnaire PNKAS-N
* Observation of clinical practice

ELIGIBILITY:
Questionnaire

Inclusion Criteria:

* nurses working at all four wards and all surgeons (experienced) at the corresponding wards

Exclusion Criteria:

* nurses not involved in clinical work

Observational study

Inclusion Criteria:

* nurses working in all four wards
* children (0-18 years) admitted to these wards during the data collection period, and their parents

Interview with children

Inclusion Criteria:

* children (6-18 years) going through surgery at all four wards during the data collection period, and their parents

Exclusion Criteria:

* children with cognitive impairment who were unable to communicate verbally
* children who did not speak Norwegian
* children younger than six years

Interview with healthcare providers

Inclusion Criteria:

* healthcare providers working in the four wards (two to four nurses, two surgeons, and two anesthesiologists in each group)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Healthcare providers' knowledge and attitudes of pediatric pain management | Baseline
  Evaluated with "The Pediatric Nurses' Knowledge and Attitudes Survey Regarding Pain Questionnaire - Norwegian version" (PNKAS-N).The questionnaire consists of 36 questions with a total score of 36. The scale ranges from minimum 0 to maximum 36 (best score).
Changes in Healthcare providers' knowledge and attitudes of pediatric pain management | short term - one month after intervention and long term - six and 12 months after intervention
  Evaluated with "The Pediatric Nurses' Knowledge and Attitudes Survey Regarding Pain Questionnaire - Norwegian version" (PNKAS-N). The questionnaire consists of 36 questions with a total score of 36. The scale ranges from minimum 0 to maximum 36 (best score).

SECONDARY OUTCOMES:
Nurses' pediatric postoperative pain management practices in surgical wards | Baseline
  Evaluated with non-participant observation using a structured observational tool (checklist) and field notes
Changes in nurses' pediatric postoperative pain management practices in surgical wards | short term - one month after intervention and long term - six and 12 months after intervention
  Evaluated with non-participant observation using a structured observational tool (checklist) and field notes
Children's experiences of pain and pain management after surgery | Baseline
  Evaluated using semi-structured face-to-face interviews with children after surgery
Healthcare providers experience barriers and facilitators for effective pediatric postoperative pain management | Baseline
  Evaluated using semi-structured focus group interviews with healthcare providers

CONTACTS AND LOCATIONS:
Overall Officials: Morten C Moe, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT03987399/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT03987399/SAP_001.pdf